CLINICAL TRIAL: NCT05527015
Title: Randomized Trial of Bifocal Spectacles vs. Single Vision Spectacles for Esotropia Greater at Near
Brief Title: Bifocal Spectacles vs. Single Vision Spectacles for Esotropia Greater at Near
Acronym: ETS3
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Concerns over recruitment feasibility
Sponsor: Jaeb Center for Health Research (Other)
Collaborators: National Eye Institute (NEI) (NIH); Pediatric Eye Disease Investigator Group (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ETS3; 2U10EY011751 (NIH)
Record Dates: First submitted 2022-08-30; First posted 2022-09-02 (Actual); Last update posted 2025-05-31 (Actual); Status verified 2025-05

CONDITIONS: Esotropia
Keywords: esotropia; bifocal
MeSH Terms: conditions — Esotropia

STUDY DESIGN:
Intervention Model Description: Random assignment (1:1) to:
  * Single vision spectacles (SVLs)
  * Bifocal spectacles (BFLs): +3.00 D flat-top 35
Who Masked: Outcomes Assessor
Masking Description: Participants will not be masked to their treatment group, given that their spectacles either will or will not have a visible flat-top bifocal. The investigator treating each participant also will not be masked to treatment group. Therefore, an examiner masked to treatment group will measure eye alignment and stereoacuity at all follow-up visits and conduct the binocular function testing at the required follow-up visits.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Single vision spectacles (SVLs) (Active Comparator)
  Interventions: Device: Single Vision Lenses
- Bifocal spectacles (BFLs) (Experimental)
  Interventions: Device: Bifocal Spectacles

INTERVENTIONS:
Device: Bifocal Spectacles — Bifocals with a +3.00 Diopter flat top 35
  Arms: Bifocal spectacles (BFLs)
Device: Single Vision Lenses — Single vision lens as prescribed by provider
  Arms: Single vision spectacles (SVLs)

SUMMARY:
Compare the proportion of BFL and SVL participants with treatment failure by 36 months, compare binocular function test scores between the BFL and SVL groups with both groups in BFL at 38 months after randomization (or 2 months after treatment failure), and evaluate treatment failure by 36 months according to baseline factor subgroups of: duration of constant esotropia pre-enrollment, presence of near stereoacuity on the Randot Preschool Stereoacuity test, in-office response of near alignment with +3.00 D lenses, and gradient AC/A ratio

DETAILED DESCRIPTION:
Participants will be randomly assigned to treatment with a BFL or SVL spectacle correction for 3 years. Generally, participants will be followed at 3-month intervals for the first year and every 6 months thereafter until the primary outcome visit at 36 months. At each follow-up visit between 3 months and 36 months, ocular alignment and stereoacuity will be assessed to determine if any of the three study-specified failure criteria have been met (worsening of distance esotropia (ET), reduction in near stereoacuity, or frequent diplopia ("more than 2 times per day" over the last week). The primary outcome is failure at or before 36 months.

If a failure criterion is met between 3 to 30 months, participants randomized to SVLs will be prescribed BFLs and those in BFLs will be prescribed continued BFLs. Participants in both groups will return in BFLs 2 months after failure for a Post-failure Secondary Outcome Visit to determine the child's binocular function, after which the child will be released to treatment at investigator discretion. Participants with confirmed failure who complete the Post-failure Secondary Outcome Exam will return for the 12- and 24-month follow-up visits (abbreviated testing) as well as the 38-month Secondary Outcome Visit (they will not return for the 36-month Primary Outcome visit).

If a failure criterion is not met between 3 to 30 months, participants without confirmed failure will complete the 36-month Primary Outcome Visit, After the 36-month visit, SVL group participants will be prescribed BFLs and BFL participants will continue using BFLs.

All participants (i.e., regardless of failure status) will return for a 38-month Secondary Outcome Visit to assess binocular function.

ELIGIBILITY:
Inclusion Criteria:

* Age 3 to <9 years
* Esodeviation meeting all the following criteria is present in refractive correction (if required or worn)

  * Constant or intermittent esotropia ≥10∆ measurable by SPCT at near
  * Distance esotropia (constant, intermittent), esophoria, or orthophoria, with near esodeviation ≥10∆ larger than distance deviation by PACT

    * If constant ET at distance, then must be ≤6∆ by SPCT
    * If intermittent ET or esophoric at distance, can be any magnitude at distance (as long as near esodeviation is ≥10∆ larger than distance deviation by PACT)
* Cycloplegic refraction within past 3 months (but not on day of exam)
* Wearing spectacles for at least 4 weeks if refractive error is 0.75 D SE or more
* Spectacles (if worn) must meet the following criteria:

  * SE refractive error must be corrected within ±0.625 D
  * Sphere power must be corrected within ±0.50 D
  * Anisometropia must be corrected within ±0.50 D SE
  * Cylinder power must be corrected within ±0.50 D
  * Cylinder axis must be within ±10 degrees if cylinder power is ≤1.00 D and within ±5 degrees if cylinder power is >1.00 D.
* Best-corrected VA meeting the following criteria:

  * Better-seeing eye VA is age-normal (see section 2.2)
  * IOD in VA within 0.2 logMAR (although previous amblyopia is allowed)
  * Worse-seeing eye VA of 20/63 or better
* Investigator and parent willing to forgo treatment of ET other than assigned randomized treatment for 36 months unless failure criteria are met.
* Investigator willing to prescribe BFL-spectacles only (in both treatment groups) for 2 months after meeting failure criteria (if failed prior to 36 months); otherwise, between 36 and 38 months

Exclusion Criteria:

* Previous BFL wear (SVL spectacle wear of any duration is allowed)
* Current or planned contact lens wear over the next 3 years
* Myopic refractive error of more than -6.00 D SE
* Previous strabismus surgery (including Botox injection), intraocular surgery (e.g., laser, anti-VEGF injection, or cataract), extraocular surgery (e.g., scleral buckle), or refractive surgery
* Previous treatment for ET using miotics, VT, or prism within prior 3 months
* Amblyopia treatment other than refractive correction within prior 3 months
* Vertical deviation ≥3Δ at distance or near by PACT
* Oculomotor findings consistent with infantile ET (e.g., latent nystagmus, manifest nystagmus, DVD)
* AV pattern: ≥10∆ difference between upgaze and downgaze by PACT at distance
* Paretic or restrictive strabismus
* Constant exotropia at near when tested through the +3.00 D add (intermittent XT and exophoria are allowed)
* Diplopia "more than 2 times per day" over the last week prior to enrollment by parental report. The frequency of diplopia, if any, must be "2 times or less per day" to be eligible.
* Significant developmental delay that would interfere with child's ability to complete testing
* Neurological conditions that could affect ocular motility (e.g., cerebral palsy, Down syndrome)
* Immediate family member (child or sibling) of any site personnel directly affiliated with the study

Ages: 3 Years to 9 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2025-09 (Estimated); Primary Completion 2033-12 (Estimated); Study Completion 2034-02 (Estimated)

PRIMARY OUTCOMES:
Number of Participants meeting treatment failure at any follow up visit before 36 months | 36 months
  Failure criteria can be described as
  1. Distance motor failure: Constant ET ≥15∆ by simultaneous prism and cover test (SPCT) at distance.
  2. Near stereo failure: Decrease in near stereoacuity on the Randot Preschool Stereotest of 2 or more levels from baseline or from 960" at baseline to nil (criteria not applicable if nil near stereo at baseline)
  3. Binocular diplopia with a frequency of "more than 2 times per day" over the last week by parental report
  4. Nonsurgical or surgical treatment for ET, other than the randomized treatment, is started before a failure criterion is met

CONTACTS AND LOCATIONS:
Overall Officials: Michael X Repka, MD, MBA, Study Chair — Wilmer Eye Institute, Johns Hopkins University

DOCUMENTS (2):
  • Study Protocol (2022-06-01): https://cdn.clinicaltrials.gov/large-docs/15/NCT05527015/Prot_000.pdf
  • Informed Consent Form (2022-08-04): https://cdn.clinicaltrials.gov/large-docs/15/NCT05527015/ICF_001.pdf